CLINICAL TRIAL: NCT00832260
Title: Influence of Atrial Pulse Width in the Behaviour of ACap™ Confirm Algorithm.
Brief Title: IES-ACap: Influence of Atrial Pulse Width in the Behaviour of ACap™ Confirm Algorithm.
Acronym: IES-ACap
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR08004ES
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Sinus Bradycardia; Sinus Node Disease; Atrio-ventricular Block
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to collect data regarding the population of patients with a pacemaker implanted.

DETAILED DESCRIPTION:
The purpose of this observational study is to collect data regarding the population of patients whit a Zephyr™ pacemaker implanted, models 5826 and 5820, and active or passive fixation leads , when the Algorithms Acap Confirm, which automatically regulates the Atrial Pulse Width, is enabled.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an indication for implantation of a dual-chamber pacemaker;
* Patient is older than 18 years of age
* Patient has signed the study specific Informed consent document.
* Primo implant.

Exclusion Criteria:

* Patient is pregnant or nursing
* Patient is less than 18 years of age
* Patient is in New York Heart Association (NYHA) class III and IV.
* Patient has a pacemaker replacement;
* Patient is unable to attend the follow-up visits;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whit a Zephyr™ pacemaker implanted, models 5826 and 5820.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Olagüe de Ros, PhD., Principal Investigator — Hospital Universitario La Fe

RESULTS

PARTICIPANT FLOW:
Groups:
- Zephyr Pacemaker: Non-randomized study. Patients with indication of a Pacemaker model Zephyr of St. Jude Medical
Period: Overall Study
Arm/Group | Zephyr Pacemaker
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zephyr Pacemaker
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients in Whom ACap™ Confirm Algorithm is Programmed Safely to ON During the First 12 Months.
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | Zephyr Pacemaker
Number analyzed (Participants) | 70
percentage of patients | 61.9

2. Secondary Outcome: Percentage of Patients in Whom ACap™ Confirm Algorithm is Recommended at a Pulse Width of 0.4 Milliseconds (ms) During All Follow-ups (Implant, Staples Removal, 3, 6, 9 and 12 Months).
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | Zephyr Pacemaker
Number analyzed (Participants) | 70
percentage of patients | 21.4

ADVERSE EVENTS:
Time Frame: 12 months
Description: Serious Adverse Events were collected
Arm/Group | Zephyr Pacemaker
Serious Adverse Events (participants affected / at risk) | 18/70
Other Adverse Events (participants affected / at risk) | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zephyr Pacemaker (N=70)
Implant of a Percutaneous transluminal coronary angioplasty (PTCA) (Cardiac disorders) | 1 (1) — On November 2009 patient was admitted into the hospital due to chest pain. Treated by Percutaneous transluminal coronary angioplasty (PTCA) On March 2010 two stents in middle descendent artery were implanted. We were aware on the 12 month follow-up.
Hemorrhoids surgery (Gastrointestinal disorders) | 1 (1) — Hemorrhoids surgery. The patient is discharged from hospital the same day (03/12/2009).
Bipolar disorder (Psychiatric disorders) | 1 (1) — Patient was admitted due to a worsening of bipolar disorder during the hospitalization. The device was implanted on the 7th May 2009. Patient was discharged on the 12th May 2009.
Seizure crisis (Psychiatric disorders) | 1 (1) — Patient was hospitalized due to seizure crisis from 21st to 28th October 2009.
Seizure crisis (Psychiatric disorders) | 1 (1) — Patient was admitted into the hospital on the 13-Apr-2009 due to seizure crisis, during the hospitalization the device was implanted on the 07-may-2009. Patient discharged on the 29-may-2009.
Myocardial infarction (Cardiac disorders) | 1 (1) — Exitus - Death due to sudden death 05-jul-2009 (Myocardial infarction)
Pyramidal Syndrome (Nervous system disorders) | 1 (1) — Patient was admitted in neurology service due to pyramidal syndrome.
Palpitations (Cardiac disorders) | 1 (1) — Patient was admitted in emergency service of another hospital on 16-jul-2009 due to palpitations.
Stent (Cardiac disorders) | 1 (1) — Patient is implanted with stent.
Thoracic pain (Cardiac disorders) | 1 (1) — Hospitalization prolonged due to thoracic pain treated with Nitroglycerin.
Transtympanic drain (Ear and labyrinth disorders) | 1 (1) — Transtympanic drain
Decrease in immunological system (Immune system disorders) | 1 (1) — Patient was hospitalized due to a decrease in immunological system.
Tracheotomy (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient was admitted in emergency service and he was made a tracheotomy.
Hernioplasty (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient was admitted in surgery service to be made a hernioplasty.
Cerebral Hemorrhage (Vascular disorders) | 1 (1) — Patient suffered a cerebral hemorrhage which caused the patient exitus.
Death (Cardiac disorders) | 1 (1) — Patient did not present at follow-up so state of event was searched. Unknown cause.
Cholangitis (Hepatobiliary disorders) | 1 (1) — Patient is committed in emergency service on 23-oct-2009 due to acute cholangitis and is discharged on 05-nov-2009. Cholecystectomy performed.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Patient is admitted at emergency service due to dyspnea.
Prostatectomy (Reproductive system and breast disorders) | 1 (1) — Patient is admitted at hospital to proceed with prostatectomy.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumothorax tension due to a secondary traumatic punction.
Atrial Flutter (Cardiac disorders) | 1 (1) — Patient is admitted in emergency service on 10-abr-2010 due to atrial flutter
Macroscopic Hematuria (Renal and urinary disorders) | 1 (2) — Macroscopic hematuria due to antiaggregants treatment
Possible strange body in a wound. (Infections and infestations) | 1 (1) — Patient was admitted in emergency service due to possible strange body in a wound.
Palpitations (Cardiac disorders) | 1 (1) — Patient is admitted in emergency service due to palpitations. Patient was discharged on the same day of admission.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less